CLINICAL TRIAL: NCT07330635
Title: Constructing a Holistic Care New Model for Chronic Wounds and Blood Circulation Detection to Enhance Home Care Quality
Brief Title: Chronic Wounds and Blood Circulation Detection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EC1130704-E
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-09

CONDITIONS: Aging; Walking, Difficulty; Chronic Limb-Threatening Ischemia; Chronic Disease
Keywords: Poor Lower Limb Circulation; Older Adults; Chronic Disease
MeSH Terms: conditions — Mobility Limitation; Chronic Limb-Threatening Ischemia; Chronic Disease

STUDY DESIGN:
Intervention Model Description: This is a three-arm parallel interventional study comparing lower limb circulation and functional performance across young adults, older adults, and older adults with poor peripheral circulation. A 12-week group-based mixed exercise intervention is applied to the older adults and circulation-deficient groups, while the young adult group serves as a reference control without intervention.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Young Adults (Reference Control) (No Intervention): Healthy young adults aged 20-35 years serving as the reference control group. Participants will not receive any intervention but will undergo the same baseline and follow-up assessments of lower limb circulation and functional performance.
- Older adults (Exercise intervention) (Experimental): Older adults aged 65 years. Participants will engage in a 12-week, group-based exercise program (3 sessions per week, 30 minutes per session) focusing on lower limb strengthening, balance, and aerobic training.
  Interventions: Behavioral: Intervention 1: Mixed exercise program; Behavioral: Intervention 2: High-intensity rowing exercise; Behavioral: Intervention 3: Vibration exercise
- Older adults with chronic disease (Exercise intervention) (Experimental): Older adults aged 65 years and above with chronic disease. Participants will engage in a 12-week exercise program (3 sessions per week, 30 minutes per session).
  Interventions: Behavioral: Intervention 1: Mixed exercise program; Behavioral: Intervention 2: High-intensity rowing exercise; Behavioral: Intervention 3: Vibration exercise

INTERVENTIONS:
Behavioral: Intervention 1: Mixed exercise program — A 12-week, group-based mixed exercise program focusing on lower limb strengthening, balance, and aerobic training (3 sessions per week, 30 minutes per session). Exercise intensity will be adjusted based on individual fitness and circulation levels.
  Other Names: Mixed exercise program
  Arms: Older adults (Exercise intervention); Older adults with chronic disease (Exercise intervention)
Behavioral: Intervention 2: High-intensity rowing exercise — A 12-week, high-intensity lower limb rowing exercise program (3 sessions per week, 30 minutes per session), with individualized intensity adjustments based on each participant's baseline
  Other Names: Lower limb rowing exercise program
  Arms: Older adults (Exercise intervention); Older adults with chronic disease (Exercise intervention)
Behavioral: Intervention 3: Vibration exercise — A 12-week, vibration exercise program (3 sessions per week, 30 minutes per session), with individualized intensity adjustments based on each participant's baseline
  Other Names: Vibration exercise program
  Arms: Older adults (Exercise intervention); Older adults with chronic disease (Exercise intervention)

SUMMARY:
Lower limb circulatory insufficiency and the associated chronic wounds are common health problems among the elderly. These issues not only affect the individual's mobility and quality of life but also potentially increase medical costs and caregiving expenses. Traditional treatment methods often employ medications to enhance blood circulation, but these clinical approaches have limited effectiveness and induce the risk of side effects. Utilizing exercise as an intervention strategy can help improve lower limb blood circulation in the elderly while reducing the side effects associated with medications. However, due to physical frailty, elderly individuals often cannot participate in high-intensity exercises to improve their circulatory performance.

Therefore, this study will develop a lower limb circulation enhancement exercise system to improve the circulatory performance in individuals with poor lower limb circulation. It will compare the effects of lower limb circulation enhancement exercise, vibration exercise, and mixed exercise on improving blood circulation and functional performance in the elderly or individuals with poor lower limb circulation.

Participants will be randomly assigned into three groups: the lower limb circulation enhancement exercise group, the vibration exercise group, and the mixed exercise group. In addition, a separate group of young adults (control group) will serve as a reference for baseline comparisons. Initially, all participants will undergo a one-time exercise test, followed by a 12-week intervention. The lower limb circulation enhancement exercise group will perform a 30-minute leg press rowing exercise three times a week, while the vibration exercise group will engage in vibration exercise at the same frequency, and the mixed exercise group will perform group-based mixed exercise training at the same frequency. The young adult control group will not receive any intervention but will undergo the same assessments.

Outcome evaluations before and after the intervention include lower limb blood perfusion monitoring, pain scales, and functional performance assessments.

ELIGIBILITY:
Inclusion Criteria:

General criteria (applied to all participants):

Willingness to participate in this study and comply with all study procedures. Able to perform basic physical activity and complete lower limb circulatory and functional assessments.

Normal cognitive function sufficient to understand instructions and provide informed consent.

Group-specific criteria:

Young Adults (Control Group):Aged 20-40 years.No known chronic diseases or peripheral circulatory disorders.Considered healthy volunteers.

Older Adults (Healthy Elderly Group):Aged 65-95 years.No major chronic diseases affecting lower limb circulation.

Older Adults with Chronic Disease (Impaired Circulation Group):Aged 65-95 years.Diagnosed with one or more conditions known to impair peripheral circulation, including but not limited to peripheral arterial disease (e.g., atherosclerosis, thromboangiitis obliterans), chronic venous insufficiency (e.g., varicose veins), diabetes mellitus, hypertension, or hyperlipidemia.

Exclusion Criteria:

Recent acute lower limb injury resulting in tissue exudation, swelling, or other conditions that prevent safe participation in the assessment or intervention procedures.

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 425 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2027-09-04 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Lower limb blood perfusion | Baseline and after 12 weeks of intervention
  Lower limb blood perfusion will be assessed using Laser Doppler Flowmetry (LDF) and Laser Speckle Contrast Imaging (LSCI).
  For LSCI, measurements will be performed at the plantar surface beneath the hallux. The protocol includes a baseline recording period, transient arterial occlusion using an ankle cuff, and post-occlusion monitoring to capture recovery and reactive changes. Skin perfusion pressure (SPP) will be derived from the LSCI signal inflection point following cuff release, expressed in millimeters of mercury (mmHg).

SECONDARY OUTCOMES:
Functional performance (Six-Minute Walk Test) | Baseline and after 12 weeks of intervention
  Walking distance covered in six minutes on a flat surface, used to assess cardiovascular endurance and functional walking capacity.
Functional performance (30-Second Sit-to-Stand Test) | Baseline and after 12 weeks of intervention
  Number of full sit-to-stand repetitions completed in 30 seconds from a standard chair without using the arms, used to evaluate lower limb strength and functional mobility.
Functional performance (10-Meter Walk Test) | Baseline and after 12 weeks of intervention
  Walking speed over a 10-meter distance at a comfortable pace, measured to assess gait performance and walking efficiency.

CONTACTS AND LOCATIONS:
Locations (1):
- National Center for Geriatrics and Welfare Research, National Health Research Institutes, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data (IPD) due to participant privacy protection and institutional policy restrictions.